CLINICAL TRIAL: NCT01833338
Title: Coronary Artery Plaque Characterisation With Non-invasive Multi-Slice Computed Tomography and Invasive Intravascular Ultrasound and Optical Coherence Tomography in Patients With Acute Coronary Syndromes Without ST-segment Elevation
Brief Title: Non-invasive and Invasive Plaque Characterisation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated based on an included stopping rule in the study protocol
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Gabija Pundziute, Principal Investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: METcUMCG 2010.266
Record Dates: First submitted 2013-03-04; First posted 2013-04-16 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Non ST Elevation Myocardial Infarction
Keywords: Non ST elevation myocardial infarction; optical coherence tomography; intravascular ultrasound; multi-slice computed tomography
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Other): There is only one arm in this study. All patients undergo MSCT, IVUS and OCT.
  Interventions: Device: Imaging

INTERVENTIONS:
Device: Imaging — All patients undergo non-invasive (MSCT) and invasive (IVUS, OCT) imaging
  Other Names: OCT: C7-XR™ OCT Intravascular Imaging System, St.Jude Medical; IVUS: Galaxy 2 IVUS Imaging System, Boston Scientific; MSCT: Dual-source CT scanner Somatom Definition, Siemens Healhtcare

SUMMARY:
The accuracy of coronary plaque characterization with Multi-slice computed tomography as compared to intravascular ultrasound and optical coherence tomography will be investigated in patients presenting with acute coronary syndrome without ST-elevation.

ELIGIBILITY:
Inclusion Criteria:

* Chest pain suggestive for myocardial ischemia for at least 30 minutes; - Electrocardiogram (ECG) with ST-segment shifts (ST-segment depression >1 mm in at least two contiguous leads or transient ST-segment elevation > 1mm with duration of < 30 min in at least two contiguous leads) and/or T-wave changes (T-wave inversion > 1.5 mm in at least three contiguous leads); - Positive hs Troponin T > 14 ng/L or positive Troponin T <0.01 µg/L - Clinical indication for invasive coronary angiography followed by PCI of the ischemia-related target lesion; - Informed consent.

Exclusion Criteria:

* Persistent ST-elevation of >1 mm in 2 or more leads; - Need for emergency invasive coronary angiography and percutaneous coronary intervention (PCI); - Need for emergency coronary artery bypass grafting; - Presence of cardiogenic shock; - Estimated glomerular filtration rate (eGFR) < 50 ml/min; - Known allergy to iodine contrast agents; - Cardiac rhythms other than sinus rhythm; - Inability to lay supine; - Inability tot sustain a breath-hold for 15 seconds; - Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Accuracy of detection of thrombus with MSCT as compared to IVUS and OCT will be investigated. | 24 hours
  All imaging methods will be performed in each patient. A 24 hour period is the maximum allowed time gap between MSCT and invasive imaging (OCT/IVUS).

SECONDARY OUTCOMES:
Accuracy of atherosclerotic plaque characterisation with MSCT as compared to IVUS and OCT will be investigated. | 24 hours
  A maximum interval of 24 hours between MSCT and IVUS/OCT is allowed in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Gabija Pundziute, MD, PhD, Principal Investigator — Department of Cardiology; Tineke Willems, MD, PhD, Principal Investigator — Department of Radiology
Locations (1):
- University Medical Center Groningen, Departments of Cardiology and Radiology, Groningen, Provincie Groningen, Netherlands